CLINICAL TRIAL: NCT02650440
Title: Robot-assisted Locomotor Training After Severe Stroke: Discrete Versus Rhythmic Movement
Brief Title: Discrete Versus Rhythmic Gait Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thais Amanda Rodrigues (Other)
Responsible Party: Sponsor-Investigator, Thais Amanda Rodrigues, Physiotherapist, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Robotics in Stroke
Record Dates: First submitted 2016-01-05; First posted 2016-01-08 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-05

CONDITIONS: Stroke; Cerebral Vascular Disorders
Keywords: robotics; locomotion; gait; walking; rehabilitation
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders | interventions — AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Novel Protocol (Experimental): Progressive decrease of speed and guidance force on robotic gait training. Initial speed is 1.4 km/h and final speed is 1.0 km/h.
  Interventions: Procedure: Novel Protocol
- Standard Protocol (Experimental): Progressive increase of speed and decrease of guidance force on robotic gait training. Initial speed is 1.4 km/h and final speed is 1.9 km/h.
  Interventions: Procedure: Standard Protocol

INTERVENTIONS:
Procedure: Novel Protocol — All subjects performed robot-assissted LT-BWST 5 times a week for 6 weeks (30 minutes of training and 15 minutes of setup). Novel (discrete) robot-assisted LT-BWST used progressive decrease in speed. Both groups started the robot-assisted LT-BWST at the same speed of 1.4km/h. The body weight support started approximately at 40% of body weight for both groups and rapidly decreased each week. The guidance force was also progressively decreased for both groups so that the exoskeleton provided the least possible assistance to the subject.
  Arms: Novel Protocol
Procedure: Standard Protocol — All subjects performed robot-assissted LT-BWST 5 times a week for 6 weeks (30 minutes of training and 15 minutes of setup). Standard (rhythmic) robot-assisted LT-BWST used progressively increased speed each week. Both groups started the robot-assisted LT-BWST at the same speed of 1.4km/h. The body weight support started approximately at 40% of body weight for both groups and rapidly decreased each week. The guidance force was also progressively decreased for both groups so that the exoskeleton provided the least possible assistance to the subject
  Arms: Standard Protocol

SUMMARY:
The objective of this study is to compare the effects of novel versus standard locomotor training using a robotic gait orthosis (LT-RGO) after stroke. The hypothesis is that the novel LT-RGO protocol, by establishing a progressive decrease in gait velocity and guidance force, may facilitate greater motor recovery compared to the use of a standard protocol.

DETAILED DESCRIPTION:
Standard (rhythmic) robot-assisted locomotor training on a bodyweight-supported treadmill (LT-BWST) used progressively increased speed each week. Novel (discrete) robot-assisted LT-BWST used progressive decrease in speed. The novel approach of slowing down the treadmill reduced momentum. If speed had been increased (standard approach), momentum would have increased (momentum = mass * velocity); and the resulting, passive propulsion of momentum would have diminished the role of cortical skills needed to plan, initiate, and overtly control gait. In sum, the novel protocol used a slower-than-standard treadmill speed in order to provide a window of time sufficient for the corticomotor system to process information, learn, and adjust its response to internal and external feedback (eg, proprioceptive input; therapist input) during robot-assisted LT-BWST.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke and image with hemiparesis left or right;
* No more that one ischemic or hemorrhagic stroke episode;
* 06 months post-stroke;
* Verified clinical stability on medical evaluation;
* Spasticity level I or II in the Ashworth scale;
* Score 1-2 in the Functional Ambulation Scale (FAC);
* Signed informed consent.

Exclusion Criteria:

* Dependence to perform activities of daily living before the stroke;
* Lack of clinical indications for exercises (such as cardiopulmonary instability and uncontrolled diabetes);
* Severe cognitive impairment;
* Serious psychiatric change that needs psychiatric care;
* Severe osteoporosis;
* Severe spasticity of the lower limbs, deformities or fixed contractures that prevent the achievement of movements;
* Lack of resistance or disabling fatigue;
* Body weight greater than 150 kg;
* Unstable angina or other untreated heart disease;
* Chronic obstructive pulmonary disease;
* Unconsolidated fractures, pressure sores;
* Other neurological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G Goroso, Doctor, Study Chair — University of Sao Paulo; Lumy Sawaki, PhD, Study Chair — University of Kentucky
Locations (1):
- Instituto de Medicina Física e Reabilitação - Lucy Montoro, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Novel Protocol | Standard Protocol
Started | 10 | 10
Completed | 10 | 8
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Novel Protocol | Standard Protocol | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants] — Population: Two individuals from Standard Protocol did not receive allocated intervention due to clinical complications.
  Participants
    number analyzed (Participants) | 10 | 08 | 18
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 9 | 5 | 14
    >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Two individuals from Standard Protocol did not receive allocated intervention due to clinical complications.
  years
    number analyzed (Participants) | 10 | 08 | 18
    (all) | 50.6 (14.4) | 59.3 (13.8) | 50.6 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two individuals from Standard Protocol did not receive allocated intervention due to clinical complications.
  Participants
    number analyzed (Participants) | 10 | 08 | 18
    Female | 6 | 4 | 10
    Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Brazil | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Functional Ambulation Scale (FAC)
Description: The Functional Ambulation Scale (FAC) assesses an individual's independence during gait and follows a six-level scale: 0 - Patient can not walk or ask for help from two or more people; 1 - Patient requires continuous support from a person who assists with weight and balance; 2 - Patient needs continuous or intermittent support from a person to help with balance and coordination; 3 - Patient required for a person without physical contact; 4 - Patient can walk independently on the floor, but requires help on stairs and ramps; 5 - Patient can walk independently.
  This study compared the gait independence by the FAC between the two Arms, after intervention as compared to baseline.
Time Frame: Baseline and 6 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Novel Protocol | Standard Protocol
Number analyzed (Participants) | 10 | 08
units on a scale | 1 [1 to 2] | 0 [0 to 1.5]

2. Secondary Outcome: Six-minute Walking Test (6MWT)
Description: Change in distance of the gait applied test after intervention as compared to baseline
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Error); unit: meters
Arm/Group | Novel Protocol | Standard Protocol
Number analyzed (Participants) | 10 | 08
meters | 25.4 (10.4) | 7.6 (14.1)

3. Secondary Outcome: Time Up and Go (TUG)
Description: This test assesses the level of mobility of the individual to measure the time spent to get up from a chair, walk a distance of 3 meters, turn around and return. This study compared the change in the time of the gait applied test after intervention as compared to baseline.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Novel Protocol | Standard Protocol
Number analyzed (Participants) | 10 | 08
seconds | -42.1 (16.4) | -11.3 (22.9)

4. Secondary Outcome: Ten-meters Walking Test (10MWT)
Description: Change in the time of the gait applied test after intervention as compared to baseline
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Novel Protocol | Standard Protocol
Number analyzed (Participants) | 10 | 08
seconds | -52.8 (27.9) | -20.3 (30.5)

5. Secondary Outcome: Lower Limbs Fugl-Meyer
Description: The Fugl Meyer Scale is a cumulative numerical scoring system that is assessed by an individual: range of motion, pain, tenderness, upper and lower extremity motor function and balance, plus coordination and speed of movement, with total 226 points. A three-point ordinal scale is applied to each item: 0 - can not be performed, 1-performed partially and 2-performed completely. For this study it was only an evaluation of motor function of the extremity of lower limbs with a total score of 0 to 34 points. The lower score indicates greater motor impairment.
  This study compared the change in motor function of lower limbs applied scale after intervention as compared to baseline
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Novel Protocol | Standard Protocol
Number analyzed (Participants) | 10 | 08
units on a scale | 2.3 (0.8) | -1.1 (2.1)

6. Secondary Outcome: Berg Scale
Description: Berg Scale is a functional scale of equilibrium performance, based on 14 common everyday items that evaluate the static and dynamic balance. The maximum scale score is 56 and each scale item has five alternatives ranging from 0 to 4 points. A score below 45 is considered a fall risk. This study comparede the change in the balance control applied scale after intervention as compared to baseline.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Novel Protocol | Standard Protocol
Number analyzed (Participants) | 10 | 08
units on a scale | 11.1 (1.6) | 6.0 (1.9)

ADVERSE EVENTS:
Time Frame: 8 weeks.
Description: Adverse events that are not Serious Adverse Events: 0
Arm/Group | Novel Protocol | Standard Protocol
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes